CLINICAL TRIAL: NCT07261579
Title: Composite Inflammatory Parameters Ratios Enforce the Role of CRP for Monitoring Ulcerative Colitis Disease Activity
Brief Title: Composite Ratios Boost CRP's Power in Monitoring Ulcerative Colitis.
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Raafat R. Mohammed, Assistant consultant of Clinical Pathology, Benha University
Other Study IDs: E/C. S/N. R14/2025
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ulcerative Colitis Patients: Patients exhibiting clinical signs suggestive of IBD were assessed for UC diagnostic criteria, and the study inclusion and exclusion standards.
  Interventions: Diagnostic Test: C-Reactive Protein measuring CRP; Diagnostic Test: CRP to Albumin Ratio

INTERVENTIONS:
Diagnostic Test: C-Reactive Protein measuring CRP — 5-ml peripheral blood samples were aseptically obtained for a complete blood count, and ELISA estimation of serum CRP
Diagnostic Test: CRP to Albumin Ratio — Serum CRP to albumin ratio (CAR) is a combination of markers for systemic inflammation and nutritional status

SUMMARY:
Inflammatory Bowel Disease (IBD) is a chronic, recurrent condition marked by disturbed levels of various hematological inflammatory cells and a deregulated immune environment. While C-reactive protein (CRP) is a key acute-phase reactant, its high levels can persist even after inflammation subsides. Other simple, cost-effective ratios, such as the Neutrophil-to-Lymphocyte Ratio (NLR), the Platelet-to-Lymphocyte Ratio (PLR), and Albumin-related ratios, also serve as promising, reproducible markers of systemic inflammation reflecting both immune status and nutrition. This study's objective is to evaluate the diagnostic performance of these various hematological inflammatory cellular components and CRP-related ratios (like the CAR) as predictors for Ulcerative Colitis (UC) disease severity, using colonoscopic and microscopic findings as the gold standard for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfilled the diagnostic criteria for UC;
* Patients were free of exclusion criteria;
* Patients who signed the written consent were enrolled in the study

Exclusion Criteria:

* Patients who was Previously diagnosed with IBD or IBS;
* Patients with recurrence of manifestations after surgical resection;
* Patients who refused to sign the participation consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consisted of all patients exhibiting clinical signs suggestive of Inflammatory Bowel Disease were assessed for Ulcerative Colitis diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
The Correlation Between Clinical and Endoscopic Diagnostic Indices and Hematologic Ratios | 45 days
  Evaluating the role of diagnostic indices (Ulcerative Colitis Disease Activity Index (UC-DAI), Simple Clinical Colitis Activity Index (SCCAI), Fecal Calprotectin (FCP) ≥150μg/ml) in active Ulcerative Colitis (UC) and their correlation with novel hematologic inflammatory markers, including Neutrophil-to-Lymphocyte Ratio (NLR), Platelet-to-Lymphocyte Ratio (PLR), Systemic Inflammatory Response Index (SIRI), Systemic Inflammation Index (SII), and the serum C-Reactive Protein (CRP)-to-Albumin Ratio (CAR).

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of medicine, Alexandria, El Alexandria, Egypt